CLINICAL TRIAL: NCT04757285
Title: Evaluation of Serum Copeptin and Psychological Stress Level Among Healthcare Providers During COVID-19 Pandemic
Brief Title: Copeptin and Psychological Stress of Medic During COVID-19 Pandemic
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, hala mourad demerdash, Consultant Clinical Pathology, Alexandria University
Other Study IDs: 0304842
Record Dates: First submitted 2021-02-06; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Psychological Stress; Hemostatic Disorder
Keywords: psychological stress; copeptin; hormones
MeSH Terms: conditions — Stress, Psychological; Hemostatic Disorders; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: 25 healthcare personnel volunteers not working in quarantine hospitals of matched age
- healthcare providers worked in Intensive Care Units: 35 physicians (28 males and 7 females) and 35 nurses (10 males and 25 females). All volunteers were in good physical health Exclusion criteria included hypertension, diabetes mellitus, obesity BMI ≥30, subjects with serum sodium ≤135 or ≥ 145 mmol /L at baseline or females receiving contraceptive pills.
  Assigned participants were clinically evaluated for as hypertension, DM, dyslipidemia, renal function.

SUMMARY:
Psychological stress (PSS) is one of the most common problems among healthcare providers during COVID-19 pandemic. PSS influences the homeostatic equilibrium of the body, involving activation of the sympathetic nervous system and hypothalamus pituitary adrenal (HPA) axis. Copeptin; C-terminal portion of Vasopressin (AVP) precursor is stable. Nevertheless, Evidence about influence of PSS on copeptin levels is lacking. The reason we are doing this research is to determine the level of psychological stress among healthcare providers exposed to at the time of work in intensive care unit (ICU) during COVID-19 pandemic; They will be appraised every assembly for psychological stress level; before start of duty shifts (first time), one week after start (second time) and two weeks after departure from shift duties in ICU (third time) for assessment of psychological stress level and stress hormones.

DETAILED DESCRIPTION:
A total of 70 healthcare personnel volunteers participated; 35 physicians and 35 nurses. All healthcare providers' volunteers are in good physical health, Exclusion criteria included hypertension, diabetes mellitus, obesity BMI ≥30, subjects with serum sodium ≤135 or ≥ 145 mmol /L at baseline or females receiving contraceptive pills.

During the research participants will answer a questionnaire as well as three blood samples are taken.

* In the first meeting, evaluation of participant general condition; determining BMI, blood pressure. Then a small amount of blood, equal to about two millimeters, will be taken from participant arm with a syringe. This blood will be tested for serum copeptin, cortisol (fasting morning sample). The investigator will ask participant few questions to evaluate the level of stress (as anxiety, insomnia, fear of infection through questionnaire)
* The second meeting, one week after work in ICU, another blood sample will be taken from participant and determine level of psychological stress.
* The third meeting, two weeks after leave from ICU participant blood sample will be taken from participant to determine stress hormones and determine level of psychological stress.

Duration

The research takes place over six months in total.

ELIGIBILITY:
Inclusion Criteria:

physicians and nurses under age of 37 years in good health

Exclusion Criteria:

* body mass index above 30
* hypertension
* Diabetes mellitus
* females receiving contraceptive pills

Ages: 24 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthcare providers worked in ICU: 35 physicians (28 males and 7 females) and 35 nurses (10 males and 25 females). Age ranged from 24 to 37 years All volunteers were in good physical health Exclusion criteria included hypertension, diabetes mellitus, obesity BMI ≥30, subjects with serum sodium ≤135 or ≥ 145 mmol /L at baseline or females receiving contraceptive pills.
  Group Information healthcare providers designated to take duty shifts at ICU in Alexandria quarantine hospitals for two weeks during COVID-19 pandemic. And a control group of healthcare providers not assigned to work in quarantine hospitals.
  First assembly one day before enrolling to work in ICU. Second assembly at the end of first week of work, third assembly two weeks after departure from work in ICU
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
evaluation of psychological stress | four weeks for each participant.
  - Primarily outcome determination of psychological stress among doctors and nurses working in ICU through a questionnaire before duty shifts [first time] and re-evaluate it after one week of work in ICU [second time], and lastly two weeks after departure from shift duties [third time].
determine stress hormones in serum cortisol and copeptin | four weeks for each participant..
  Second to determine stress hormones copeptin and cortisol (possible stress biomarkers) concurrently with questionnaire.

SECONDARY OUTCOMES:
correlation of psychological stress with stress hormone copeptin | four weeks for each participant..
  correlate the level of psychological stress calculated from provided questionnaire in the three assemblies with stress biomarkers copeptin and cortisol in the three measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McEwen BS. Protective and damaging effects of stress mediators: central role of the brain. Dialogues Clin Neurosci. 2006;8(4):367-81. doi: 10.31887/DCNS.2006.8.4/bmcewen. PMID 17290796
- [Result] Christ-Crain M, Fenske W. Copeptin in the diagnosis of vasopressin-dependent disorders of fluid homeostasis. Nat Rev Endocrinol. 2016 Mar;12(3):168-76. doi: 10.1038/nrendo.2015.224. Epub 2016 Jan 22. PMID 26794439

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT04757285/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT04757285/ICF_001.pdf